CLINICAL TRIAL: NCT00004331
Title: Studies in Porphyria I: Characterization of Enzyme Defects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Other Study IDs: 199/11888; UTMB-399
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Porphyria
Keywords: inborn errors of metabolism; porphyria; rare disease
MeSH Terms: conditions — Porphyrias; Metabolism, Inborn Errors; Rare Diseases

SUMMARY:
OBJECTIVES: I. Characterize enzyme defects in patients with known or suspected porphyria and their family members.

II. Determine whether selected patients are eligible for other porphyria research protocols.

III. Provide blood, urine, and fecal samples from well characterized patients and their family members to investigators studying the nature of specific mutations in genes for heme biosynthetic pathway enzymes.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: All patients are evaluated for porphyria type and factors contributing to the clinical expression of their particular form of the disease. Testing includes erythrocyte porphobilinogen deaminase, erythrocyte protoporphyrin, plasma porphyrins, and urinary and fecal porphyrins and precursors.

Selected patients are entered into other porphyrin research protocols in this and other institutions, including analysis of DNA to identify specific mutations in genes for heme biosynthetic pathway enzymes.

ELIGIBILITY:
* Suspected or confirmed porphyria
* Adults, children, and family members eligible

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1992-11

CONTACTS AND LOCATIONS:
Overall Officials: Karl Elmo Anderson, Study Chair — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States